CLINICAL TRIAL: NCT00590278
Title: A Phase-II Study Of TOMUDEX Plus Radiotherapy In Subject With Inoperable or Recurrent Rectal Cancer
Acronym: TOMUDEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Tayfun Hancilar, AstraZeneca Turkey Clinical Study Information
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1694TR/01
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Inoperable or Recurrent Rectal Cancer
Keywords: Tomudex; inoperable rectal cancer; recurrent rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — raltitrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tomudex
Procedure: Radiotherapy
Procedure: Haematology
Procedure: Biochemistry

SUMMARY:
The pilot study is designed to investigate the value of Neo-adjuvant Tomudez in combination with radiotherapy in patients with inoperable or recurrent rectal cancer in terms of response rate and increasing the resectability of initially inoperable rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of inoperable/recurrent rectal cancer
* Age > 18 years
* At least 1 measurable lesion should be present
* WHO performance score < 2
* Life expentancy of at least 12 weeks
* Subjects will be considered appropriate to receive systemic chemotherapy and pelvic radiotherapy
* Documented informed consent to participate in the trial

Exclusion Criteria:

* Previous systemic chemotherapy
* Previous radiotherapy to the planned exposure area
* Subjects with distant metastases
* (a)white blood cell < 4.0x109/L (unless absolute neutrophil count is >2.0x109/L or (b) Platelet count < 100x109/L
* Serum creatinine above the upper limit of the normal range
* (a) Serum bilirubin > 1.25 times the upper limit of the normal range or (b) Asparate aminotransferase(AST) or Alanine amiontransferase (ALT) >2.5 times the upper limit of the normal range
* Any severe concurrent medical condition which would make it undesirable, in the clinician's opinion, for the patient to participate in the trial or which would jeopardise compliance with the trial period
* Pregnancy or breast feeding. Women of childbearing age must use effective contraception
* Previous or current malignancies at other sites, with the exception of adequately treated in-situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin
* Patient participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2002-08

PRIMARY OUTCOMES:
This study will evaluate the value of TOMUDEX in combination with a 'standard' course of pelvic radiotherapy for inoperable/recurrent rectal cancer, in terms of response rate and increasing the resectability rate

CONTACTS AND LOCATIONS:
Overall Officials: Tayfun Hancilar, MD, Principal Investigator — Okmeydani Hospital Istanbul
Locations (1):
- Research Site, Istanbul, Turkey (Türkiye)